CLINICAL TRIAL: NCT00657891
Title: The Effect of Xolair (Omalizumab) on Inhibiting Leukotriene and Cytokine (IL-4 and IL-13) Release From Blood Basophils
Brief Title: The Effect of Xolair (Omalizumab) on Allergy Blood Cells
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IgE 025 US22
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: Allergic Asthma; Anti IgE; Xolair; Basophil; IL-13; IL-4; Histamine
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo Injection
  Interventions: Drug: Placebo
- 2 (Experimental): Xolair at 0.016 mg/kg/IgE(iu/ml)/4 wks
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — 0.016 mg/kg/IgE(iU/ml)/4 wks, Subcutaneously
  Other Names: Xolair; rhumabe35
  Arms: 2
Drug: Placebo — Placebo Injection
  Arms: 1

SUMMARY:
We are studying Xolair (omalizumab) to see it's effect on allergic blood cells. The blood tests will be done in a test tube to see if they react differently before and after treatment. The blood cells will be mixed with to whatever the person is allergic.

DETAILED DESCRIPTION:
Must be allergic-asthma with IgE between 30 and 700 IU/ml.

ELIGIBILITY:
Inclusion Criteria:

* 2 year history of ragweed allergic rhinitis
* positive skin prick tests to ragweed >5 mm wheal diameter
* serum IgE <700 iU/m

Exclusion Criteria:

* Use of prohibited medications (e.g. antihistamine in past 7 days and topical or oral corticosteroids in past 1 month, beta-agonist or theophylline for 1 week
* History of immunotherapy in the past 2 years
* Exposure to Omalizumab in the past 2 years
* Clinically significant non-allergic or perennial rhinitis to avoid mediator release due to environmental allergens
* Asthma other than mild intermittent
* Women of childbearing potential who are not on an accepted form of birth control, as well as women who are breastfeeding
* Known sensitivity to study drug Xolair
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Patients with a previous history of cancer
* Use of any other investigational agent in the last 30 days

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine if Xolair (omalizumab) inhibits basophil leukotriene secretion & to compare this with its inhibition of histamine release. We will also compare this inhibition in basophils stimulated with allergen vs anti-IgE vs calcium ionophore. | 1 year

SECONDARY OUTCOMES:
To determine the effect of Xolair (omalizumab) on IL-4 &vIL-13 secretion. To compare the effect of Xolair on IL-4 vs IL-13 secretion from basophils stimulated with allergen, anti-IgE & calcium ionophore (ionomycin). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Townley, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States